CLINICAL TRIAL: NCT01690780
Title: Oral Morphine Versus Ibuprofen for Post-fracture Pain Management in Children: a Randomized Controlled Study
Brief Title: Oral Morphine Versus Ibuprofen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Naveen Poonai (Other)
Responsible Party: Sponsor-Investigator, Naveen Poonai, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-11-340; 18091 (Other: REB)
Record Dates: First submitted 2012-09-13; First posted 2012-09-24 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Upper Extremity Fractures; Analgesia Post Fracture
Keywords: fracture; pediatric; oral morphine; ibuprofen
MeSH Terms: conditions — Fractures, Bone | interventions — Morphine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen
- Oral morphine (Experimental)
  Interventions: Drug: Oral morphine

INTERVENTIONS:
Drug: Oral morphine — oral morphine 0.5 mg/kg (max 10 mg) every 6 hours as needed for 24 hours
  Arms: Oral morphine
Drug: Ibuprofen — Ibuprofen 10 mg/kg (max 600 mg) every 6 hours as needed for pain (maximum 4 doses) for 24 hours following discharge from the emergency department
  Arms: Ibuprofen

SUMMARY:
Children 5-17 years of age who have sustained a non-operative distal forearm (radius and/or ulna) or clavicular fracture will be randomized to receive either ibuprofen or oral morphine as needed for pain relief for the first 24 hours following discharge from the emergency department. Pain will be assessed using the self-report Faces pain scale revised (FPS-R). We hypothesize that oral morphine will result in greater pain relief than ibuprofen.

ELIGIBILITY:
Exclusion Criteria:

* patients with known hypersensitivity to either ibuprofen or morphine
* chronic users of NSAIDS or opioids
* fractures requiring operative management
* associated injuries requiring analgesia
* poor English fluency
* pregnancy

Inclusion Criteria:

* All patients aged 5 to 17 years with a non-operative forearm or distal radius fracture

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 183 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Faces Pain scale - revised | 30 minutes post intervention compared to baseline
  The primary outcome variable is the pre-post intervention difference in pain scores as measured by self-reported Faces Pain Scale - Revised (FPS-R) for the first 24 hours post-fracture management following the as needed administration of the study drugs.

SECONDARY OUTCOMES:
Acetaminophen doses | 24 hours
  The secondary outcome variable is the number of breakthrough acetaminophen doses required/taken by the participant for the first 24 hours post-fracture management

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Poonai, MD, FRCPC, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

REFERENCES:
- [Derived] Faught L, Elzagallaai AA, Tonial N, Ali S, Lepore N, Reardon J, Urquhart B, Ross C, Rieder MJ, Poonai N. Oral morphine pharmacokinetics in healthy children and the effect of genetic polymorphisms: An exploratory study. Paediatr Child Health. 2025 Oct 12;31(1):35-41. doi: 10.1093/pch/pxaf084. eCollection 2026 Feb. PMID 41630937
- [Derived] Poonai N, Bhullar G, Lin K, Papini A, Mainprize D, Howard J, Teefy J, Bale M, Langford C, Lim R, Stitt L, Rieder MJ, Ali S. Oral administration of morphine versus ibuprofen to manage postfracture pain in children: a randomized trial. CMAJ. 2014 Dec 9;186(18):1358-63. doi: 10.1503/cmaj.140907. Epub 2014 Oct 27. PMID 25349008